CLINICAL TRIAL: NCT04587414
Title: Personalized eHealth Intervention in Patients With Type 2 Diabetes to Promote Daily Physical Activity Utilizing 24h Self-monitoring - Implementation Frustrated by COVID-19 Epidemic
Brief Title: eHealth Intervention on Physical Activity for Type 2 Diabetics - Frustrated by COVID-19
Acronym: MySteps-CoV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UKK Institute (Other)
Collaborators: North Karelia Hospital District (Unknown); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Harri Sievanen, Research Director, UKK Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MySteps ETL 303/2017
Record Dates: First submitted 2020-09-08; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Type2 Diabetes
Keywords: physical activity; sedentary behavior; accelerometer; eHealth; COVID-19
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; COVID-19 | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The study is a pragmatic three-arm randomized controlled trial carried out within the primary health care setting. Besides the usual care given to type 2 diabetics, the patients may be assigned either into a 6-month eHealth intervention complemented by face-to-face and telephone counselling contacts on physical activity or into a 6-month eHealth intervention without counselling contacts. After the 6-month intervention, there is a 6-month follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eHealth + counselling contacts (Experimental): 6-month eHealth physical activity intervention complemented by face-to-face and telephone counselling contacts on physical activity..
  Interventions: Behavioral: eHealth +counselling contacts; Behavioral: Usual care
- eHealth (Experimental): 6-month eHealth physical activity intervention
  Interventions: Behavioral: eHealth; Behavioral: Usual care
- Usual care (Other): Usual care of type 2 diabetics within the primary health care setting.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: eHealth +counselling contacts — The 6 month eHealth intervention comprises continuous self-monitoring of PA and SB using hip-worn accelerometer and ExSed application, which gives cloud-computed personal feedback about accelerometer-measured PA and SB on smartphone and provides a platform for a health care professional to set and monitor patient's personal activity goals as well as give personalized feedback to the patient. In addition, instructions and video-demonstrations on how to reach the goals are provided via Internet. The eHealth intervention is complemented by face-to-face and telephone counselling on physical activity which comprises 4 to 6 contacts between a health care professional and the patient as well as at least 3 telephone contacts during 6 months.
  Arms: eHealth + counselling contacts
Behavioral: eHealth — The 6 month eHealth intervention comprises continuous self-monitoring of PA and SB using hip-worn accelerometer and ExSed application, which gives cloud-computed personal feedback about accelerometer-measured PA and SB on smartphone and provides a platform for a health care professional to set and monitor patient's personal activity goals as well as give personalized feedback to the patient. In addition, instructions and video-demonstrations on how to reach the goals are provided via Internet. No telephone calls nor face-to-face counselling contacts on physical activity are taken.
  Arms: eHealth
Behavioral: Usual care — Usual care and councelling given to type 2 diabetics within the primary health care setting.

SUMMARY:
This pragmatic 3-arm randomized controlled trial is conducted within the primary health care setting. The trial evaluates the effectiveness of a personalized eHealth intervention based on a hip-worn accelerometer, smartphone application and cloud service (www.exced.com) with or without face-to-face and telephone counselling contacts on physical activity (PA) compared to usual care in increasing daily PA and reducing sedentary behavior (SB) among type 2 diabetes (T2D) patients.The duration of the intervention period is 6 months, after which there is a 6 month follow-up for evaluating the maintenance of anticipated intervention effects. The primary goal of the intervention is that the T2D patients increase their daily number of steps by replacing SB with low intensity PA. The secondary goal is to increase short bouts of moderate-to-vigorous PA according to personal goals. It is expected that the eHealth intervention complemented by individual counselling is the most effective in reaching the goals, and the eHealth intervention is more effective than usual care.

Measurements are done at baseline, after the 6-month intervention, and after the 6-month follow-up. Participants' one-week PA and SB are measured with a hip-worn triaxial accelerometer and analyzed with validated algorithms. Cardiorespiratory fitness is assessed with a validated 6-minute walk test. Diabetes-related metabolic biomarkers (HbA1C, LDL-c, HDL-c, oxidized LDL and HDL lipids) and cardiovascular risk factors (blood pressure, BMI, waist circumference) are measured with standard laboratory methods. Quality of life is assessed by RAND-36 method. The interventions are evaluated with RE-AIM (Reach, Effectiveness, Adoption, Implementation and Maintenance) method. Besides effectiveness, RE-AIM methods evaluates the target group reach and adherence; provider adoption; intervention fidelity; maintenance of the changes in PA and SB behavior, biomarkers and CVD risk factors; intervention transferability to clinical practice; adverse events; and patient and provider satisfaction.

Unexpectedly, the COVID-19 pandemic in spring 2020 led to substantial restrictions in outdoors mobility of T2D patients and their access access to health care in Finland, facts that frustrated the planned implementation of the original intervention, related measurements and their scheduling. This means that not all planned measurements could be done at all or at the scheduled time point. Irrespective of the time of recruitment, all follow-up measurements are done from June to September 2020. Notwithstanding the COVID-19 pandemic annulled the original intervention, the collected data yet provides unique insights into measured physical activity, fitness and metabolic biomarkers of T2D patients before and during the COVID-19 pandemic and consequent restrictions.In addition, the data allows to evaluate the implementation of eHealth approach and face-to-face and telephone PA counselling contacts within the primary health care setting.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosed type 2 diabetes
* a prescheduled appointment with a health care professional regarding PA counselling in primary care settings of North Karelia Hospital District, Finland
* body mass index <40
* does not meet the current PA recommendation for health
* is able to conduct six minute walk test.

Exclusion Criteria:

* any problem that limits ability to walk without an aid
* any health problem that hinders participation in light to moderate intensity PA,
* not able or willing to use smartphone
* not willing to wear the research accelerometer at the baseline

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in total mean daily step count | At 6 and 12 months compared to baseline (0 months). N.B. Because of COVID-19, the schedule and contents of measurements may change individually depending on the time of recruitment.
  Step count during one week is measured with a hip-worn accelerometer at baseline, 6 months, and 12 months

SECONDARY OUTCOMES:
Changes in total mean daily time of sedentary, low intensity PA and moderate-to-vigorous PA | at 6 and 12 months compared to baseline (0 months). N.B. Because of COVID-19, the schedule and contents of measurements may change individually depending on the time of recruitment.
  Sedentary time and PA time at different intensity ranges are measured with a hip-worn accelerometer at baseline, 6 months and 12 months
Changes in the mean daily number of moderate-to-vigorous PA bouts lasting at least 1, 5 and 10 minutes. | at 6 and 12 months compared to baseline (0 months). N.B. Because of COVID-19, the schedule and contents of measurements may change individually depending on the time of recruitment.
  Durations of moderate-to-vigorous PA bouts measured with a hip-worn accelerometer at baseline, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tommi Vasankari, MD, PhD, Principal Investigator — UKK Institute
Locations (1):
- North Karelia Hospital District, Joensuu, Finland

IPD SHARING:
Plan to Share IPD: No